CLINICAL TRIAL: NCT06463353
Title: A Multicenter, Randomized, Double-blind, Controlled Clinical Study of Xia's Dermatology Method of Nourishing Blood and Moistening Dryness to Prevent Relapse in Remission of Moderate-to-severe Atopic Dermatitis
Brief Title: Clinical Study of Trilinolein Cream for Prevention of Relapse in Remission of Moderate-to-severe Atopic Dermatitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Yueyang Integrated Medicine Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-134
Record Dates: First submitted 2024-06-06; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trilinolein cream group (Experimental): receiving trilinolein cream twice a day,in the morning and evening, for a period of 12 weeks.
  Interventions: Other: trilinolein cream group
- cream base group (Placebo Comparator): receiving cream base twice a day,in the morning and evening, for a period of 12 weeks.
  Interventions: Other: cream base group

INTERVENTIONS:
Other: trilinolein cream group — Apply trilinolein cream evenly to the affected skin twice daily. The dosage is calculated using Finger Tip Units (FTU) and should not exceed a maximum of 30 grams per day.
  Arms: Trilinolein cream group
Other: cream base group — Apply cream base evenly to the affected skin twice daily. The dosage is calculated using Finger Tip Units (FTU) and should not exceed a maximum of 30 grams per day.
  Arms: cream base group

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled will be conducted at Yueyang Hospital of Integrative Medicine, Shanghai University of Traditional Chinese Medicine; Seventh People's Hospital, Shanghai University of Traditional Chinese Medicine; Jiading District Hospital of Traditional Chinese Medicine, Shanghai; and Baoshan District Hospital of Integrative Medicine, Shanghai; Huashan Hospital affiliated with Fudan University, Longhua Hospital affiliated with Shanghai University of Traditional Chinese Medicine, Shuguang Hospital affiliated with Shanghai University of Traditional Chinese Medicine, and the First Affiliated Hospital of the Naval Medical University. Approximately 376 participants will be recruited and randomly assigned to the Trilinolein cream or cream base group using block group randomization. The primary outcome will be time to relapse (number of days from the start of dosing to the time of relapse rating), and secondary outcomes will include eczema area and severity indices, overall investigator ratings, visual itch analog scores, dermatologic quality of life indices, overall improvement rates, and safety metrics. All data from the study will be analyzed using the SPSS 23.0 statistical package.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled trial will be conducted at Huashan Hospital affiliated with Fudan University, Longhua Hospital affiliated with Shanghai University of Traditional Chinese Medicine, Shuguang Hospital affiliated with Shanghai University of Traditional Chinese Medicine, the First Affiliated Hospital of Naval Military Medical University, Yueyang Hospital of Traditional Chinese Medicine and Western Combined Hospital affiliated with Shanghai University of Traditional Chinese Medicine, the Seventh People's Hospital affiliated with Shanghai University of Traditional Chinese Medicine, Shanghai Jiading Hospital of Traditional Chinese Medicine, and the Combined Hospital of Traditional Chinese Medicine and Western Combined Hospital of Baoshan District of Shanghai. . The trial will start after ethical approval and protocol registration. Patient recruitment started in June 20234 and is expected to end in March 20257 . It is anticipated that 376 participants will be enrolled in the trial and randomly assigned in a 1:1 ratio to receive treatment with Trilinolein cream or cream base. The Standards for Reporting Interventions in Acupuncture Clinical Trials (STRICTA) and the SPIRIT Reporting Guidelines will be followed in the development of the standard protocol to clearly and transparently explain the relevant treatment processes.

Potential subjects will be evaluated for eligibility to determine if inclusion and exclusion criteria are met. Eligible subjects will voluntarily provide written informed consent prior to randomization.

The study will have a double-blind design.Trilinolein cream and cream base will be supplied by the manufacturer, registered, and then distributed by the designated investigator at the time of the visit. Unused cream will be collected and counted after each distribution except for the first distribution.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a clear diagnosis of atopic dermatitis in accordance with the diagnostic criteria of Chinese and Western medicine;
2. Age ≥2 years and ≤75 years; gender is not limited;
3. Patients with a previous history of moderate to severe atopic dermatitis (EASI score ≥ 8, or SCORAD score ≥ 26, or IGA score ≥ 3);
4. Patients were in AD remission with a skin lesion IGA score ≤ 1 for 2 consecutive weeks;
5. All patients or guardians signed an informed consent form, of which the guardian signed the informed consent form for patients aged 2-8 years (<8); the patient and guardian signed the informed consent form for patients aged 8-18 years (<18); and the patient signed the informed consent form for patients aged 18-75 years.

Exclusion Criteria:

1. Patients who are in the acute morbid stage and have erosion, exudation, and secondary infection;
2. Patients who are allergic to the test article and its components;
3. Patients who are currently participating in other clinical studies or have participated in other clinical studies within 1 month;
4. Patients with skin diseases other than AD in the area to be treated;
5. Patients with severe hepatic or renal diseases, hematologic disorders, autoimmune diseases, chronic severe infections, diabetes or diseases of God, drug or alcohol abuse;
6. Suffering from malignant tumors or other serious diseases that may affect the correct assessment of efficacy;
7. Have been treated with dupliyuzumab with a discontinuation time ≤ 12 weeks, or have been treated with a JAK inhibitor with a discontinuation time ≤ 1 week;
8. Patients who have been systematically treated with hormones, other immunosuppressive agents (cyclosporine, methotrexate, reglanoside, etc.) or phototherapy;
9. Other reasons (e.g., poor compliance, inability to follow up as scheduled) that the investigator believes preclude enrollment.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 376 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence time | Assessed at screening period -14 ~ -1 days (V1), treatment period day 1 (V2), week 4 ± 3 days (V3), week 8 ± 3 days (V4), week 12 ± 3 days (V5) and follow-up period week 16 ± 3 days (V6)
  number of days from start of dosing to time of relapse assessment

SECONDARY OUTCOMES:
Eczema Area and Severity Index(EASI) | Assessed at screening period -14 ~ -1 days (V1), treatment period day 1 (V2), week 4 ± 3 days (V3), week 8 ± 3 days (V4), week 12 ± 3 days (V5) and follow-up period week 16 ± 3 days (V6)
  One of the commonly used assessment indicators for atopic dermatitis
Investigator's Global Assessment(IGA) | Assessed at screening period -14 ~ -1 days (V1), treatment period day 1 (V2), week 4 ± 3 days (V3), week 8 ± 3 days (V4), week 12 ± 3 days (V5) and follow-up period week 16 ± 3 days (V6)
  One of the commonly used assessment indicators for atopic dermatitis
Visual Analogue Scale(VAS) | Assessed at screening period -14 ~ -1 days (V1), treatment period day 1 (V2), week 4 ± 3 days (V3), week 8 ± 3 days (V4), week 12 ± 3 days (V5) and follow-up period week 16 ± 3 days (V6)
  One of the commonly used assessment indicators for atopic dermatitis
Dermatology Life Quality Index(DLQI) | Assessed at screening period -14 ~ -1 days (V1), treatment period day 1 (V2), week 4 ± 3 days (V3), week 8 ± 3 days (V4), week 12 ± 3 days (V5) and follow-up period week 16 ± 3 days (V6)
  One of the commonly used assessment indicators for atopic dermatitis
Overall effective rate | through study completion, an average of 16 weeks
  Difference between pre- and post-treatment EASI scores/baseline EASI score × 100%, where ≥90% is considered cured, 60% ~ 89% is considered effective, 20% ~ 59% is considered improved, and <20% is considered ineffective, and the total of the cured rate and the effective rate is the overall effective rate.
Total serum IgE | Assessed at screening period -14 ~ -1 days (V1), treatment period week 4 ± 3 days (V3), week 12 ± 3 days (V5)
  Peripheral blood samples are collected from patients by sub-centers and uniformly sent for testing by the main center.
Trans Epidermal Water Loss(TEWL) | Assessed at screening period -14 ~ -1 days (V1), treatment period day 1 (V2), week 4 ± 3 days (V3), week 8 ± 3 days (V4), week 12 ± 3 days (V5) and follow-up period week 16 ± 3 days (V6)
  Indicators for objective evaluation of treatment
Skin flora test | Assessed at treatment period day 1 (V2) and follow-up period week 16 ± 3 days (V6)
  Detecting changes in flora species and diversity
Safety evaluation indicators | up to 12 weeks
  Record adverse events in detail at any time, and record any adverse reactions such as hyperpigmentation, capillary dilatation and skin atrophy at the site of application during the period of drug administration